CLINICAL TRIAL: NCT05115227
Title: Long-term Multidisciplinary Team-based Management of Back Pain: Development and Feasibility (TeamBack Trial)
Brief Title: Long-term Multidisciplinary Team-based Management of Back Pain
Acronym: TeamBack
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spine Centre of Southern Denmark (Other)
Collaborators: Department of Sports Science and Clinical Biomechanics, University of Southern Denmark (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TeamBack
Record Dates: First submitted 2021-10-13; First posted 2021-11-10 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Educational Status; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multidisciplinary (Experimental): A pragmatic team-based management approach is individualized for each patient.
  Interventions: Behavioral: Education; Behavioral: Exercise

INTERVENTIONS:
Behavioral: Education — The team will educate the patient about low back pain and how this can be self-managed.
  Other Names: Long-term team-based support
Behavioral: Exercise — The team will advice the patient to conduct relevant exercises and to stay physical active.

SUMMARY:
Long-term approaches are challenging to implement within the current care system, which rewards clinicians for attempting to quick-fix a long-term condition. This results in increased inappropriate imaging, opioid prescriptions, surgery, and visits/rehabilitation in secondary care, leading to higher societal costs and the continuing increase of LBP-related disability that is currently observed.

The investigators argue that LBP management can be optimized by providing patients with self-management strategies supported by a multidisciplinary team and providing simple, safe, and low-cost interventions that adhere to clinical guidelines. This has the potential to change patient behaviors and facilitate empowerment to self-manage LBP leading to lower societal costs of LBP.

Research objectives

The investigators will develop and test a long-term supportive multidisciplinary team-based management strategy with a specific focus on communicating a structured and unchanging message about individualized diagnosis, treatment, and prognosis, focusing on conducting a large randomized controlled trial as the next phase.

This feasibility trial will be completed in a secondary care settings, where relevant patients with poor management skills and insufficient effects of usual (primary) care management can be identified.

The specific objectives are:

(I) To develop a long-term supportive multidisciplinary team-based management strategy for secondary-care low back pain patients

(II) To test the feasibility by assessing:

* Changes in relevant outcomes
* Utilization of Primary care
* Patients and clinicians experience with the intervention
* Practical challenges of the setting

The management strategy development follows the principles provided by the Medical Research Council for developing complex interventions.

Development of the framework

Step 1: Framework setup

The investigators constructed a basic framework for the intervention by reviewing relevant systematic reviews and clinical guidelines. The research group determined the initial management intervention. Afterward, the investigators conducted a small survey on 191 participants (11% of the total sample of patients between February and May 2021), about their interest in participating. The majority would find such an approach of interest (147(77%)). In parallel, the investigators conducted short semi-structured interviews concerning the intervention with a convenient sample of 20 patients. Seventeen provided usable data.

Step 2 - Development

Using the participants' information, the investigators re-framed the management strategy. Subsequent semi-structured focus-group interviews with a clinical panel for further modifications before testing was conducted.

Step 3 - Feasibility

The multidisciplinary team for the feasibility trial consists of two coordinators (chiropractors), two therapists (physical therapists), one medical doctor, and one nurse.

The feasibility trial aims to identify and develop the appropriate framework by:

I) Investigating the patients' experiences of the current management strategy II) Ensuring satisfactory work-relations between clinicians III) Determining the primary outcome IV) Mapping the multiple interacting components of the management strategy V) Investigating how to measure parallel use of primary care and how this could be applied in the trial evaluation VI) Estimating the workload (number of hours) of the clinicians VII) Quantifying any out-of-protocol behaviors by clinicians and patients alike VIII) Quantifying the different aspects of the intervention using the clinical records

The feasibility trial will include 25 LBP patients from the Spine Centre willing to participate in a limited three-month follow-up.

The intervention procedure is:

1) A team meeting will be held each morning where the coordinator and the feasibility team will go through the patients. This will start the initial sparring process to ensure a structured and unchanging message for the patient.

The coordinator will first assess each patient face-to-face according to ICD-10 principles and enroll eligible patients in the trial. Afterward, the therapist will evaluate the patient's current functional status and management strategy. During the three months, patients will have multiple encounters with the coordinator, the therapist, and the nurse, if needed. The therapist will provide further interventions (e.g., exercise and cognitive/behavioral therapy) to encourage self-management.

The investigators will assess the following outcomes at three months: Disability (primary), pain, self-efficacy, quality of life, LBP trajectory, workability, and work retention.

ELIGIBILITY:
Inclusion Criteria:

* Able to speak Danish
* Disability score > 40%
* Duration of current episode > 3 months

Exclusion Criteria:

* Surgical candidate due to acute radiculopathy
* Malignant or inflammatory back pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-11-10 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2022-04-20 (Actual)

PRIMARY OUTCOMES:
Disability | Changes in mean values from baseline to 3 months
  The Oswestry disability index

CONTACTS AND LOCATIONS:
Overall Officials: Casper G Nim, PhD, Principal Investigator — Spine Center of Southern Denmark, University Hospital of Southern Denmark
Locations (1):
- Spine Centre of Southern Denmark, Middelfart, Denmark

IPD SHARING:
Plan to Share IPD: No
We have no plans of sharing the individual participant data, as there is no available data for secondary analyses.